CLINICAL TRIAL: NCT04489381
Title: Phase 3, A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Efficacy and Safety of Nitazoxanide in the Treatment of Colds Due to Enterovirus/Rhinovirus Infection
Brief Title: Trial to Evaluate Efficacy and Safety of Nitazoxanide in the Treatment of Colds Due to Enterovirus/Rhinovirus Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM08-3009
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Enterovirus; Rhinovirus
Keywords: Enterovirus; Rhinovirus
MeSH Terms: conditions — Enterovirus Infections | interventions — nitazoxanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitazoxanide (Active Comparator): Two nitazoxanide 300 mg tablets orally twice daily for 5 days
  Interventions: Drug: Nitazoxanide; Dietary Supplement: Vitamin Super B-Complex
- Placebo (Placebo Comparator): Two placebo tablets orally twice daily for 5 days
  Interventions: Drug: Placebo; Dietary Supplement: Vitamin Super B-Complex

INTERVENTIONS:
Drug: Nitazoxanide — Two nitazoxanide 300 mg tablets administered orally twice daily with food for 5 days
  Other Names: NTZ (nitazoxanide); NT-300
  Arms: Nitazoxanide
Drug: Placebo — Two placebo tablets administered orally twice daily with food for 5 days
  Arms: Placebo
Dietary Supplement: Vitamin Super B-Complex — Vitamin Super B-Complex administered orally twice daily to maintain the blind

SUMMARY:
Trial to evaluate the efficacy and safety of nitazoxanide in the treatment of colds due to enterovirus/rhinovirus infection

DETAILED DESCRIPTION:
Multicenter, randomized, double-blind trial to evaluate the efficacy and safety of nitazoxanide in the treatment of colds due to enterovirus/rhinovirus infection

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 12 years of age
* Presence of clinical signs and/or symptoms consistent with worsening or stable cold due to Enterovirus/Rhinovirus infection (one of the following is required):

  1. Presence of at least two respiratory symptom domains (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO OR
  2. Presence of at least one respiratory symptom domain (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO with pulse rate ≥90 OR
  3. Presence of at least one respiratory symptom domain (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO with respiratory rate ≥16

AND patient reported assessment that symptoms are present, the symptoms are not consistent with the subject's usual health, the symptoms interfere with daily activities, and the symptoms have worsened or remained the same relative to the previous day, as confirmed by responses to questions in the Screening FLU-PRO.

* Onset of symptoms no more than 72 hours before enrollment in the trial. Onset of symptoms is defined as the earlier of the first time at which the subject experienced subjective fever or any respiratory symptom (head, throat, nose, chest, or cough symptoms).
* Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of the subject diary and all protocol procedures.

Exclusion Criteria:

* Subjects who experienced a previous episode of acute upper respiratory tract infection, otitis, bronchitis or sinusitis or received antibiotics for these conditions within two weeks prior to and including study day 1.
* Severely immunodeficient persons including:

  1. Subjects with immunologic disorders or receiving immunosuppressive therapy (e.g., for organ or bone marrow transplants, immunomodulatory therapies for certain autoimmune diseases).
  2. Subjects with untreated human immunodeficiency viruses (HIV) infection or treated human immunodeficiency viruses (HIV) infection with a CD4 count below 350 cells/mm3 in the last six months.
  3. Subjects actively undergoing systemic chemotherapy or radiotherapy treatment for malignancy.
  4. Subjects using steroids as maintenance therapy for a chronic condition.
* Subjects with active respiratory allergies or subjects expected to require anti- allergy medications during the study period for respiratory allergies.
* Females of childbearing potential who are either pregnant or sexually active without the use of birth control. Female subjects of child-bearing potential that are sexually active must have a negative baseline pregnancy test and must agree to continue an acceptable method of birth control for the duration of the study and for 1 month post-treatment. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an Intrauterine Device (IUD), or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. Female subjects are considered of childbearing potential unless they are postmenopausal (absence of menstrual bleeding for 1 year - or 6 months if laboratory confirmation of hormonal status), or have had a hysterectomy, bilateral tubular ligation or bilateral oophorectomy.
* Subjects residing in the same household with another subject participating in the study.
* Treatment with any investigational drug or vaccine therapy within 30 days prior to screening and willing to avoid them during the course of the study.
* Receipt of any dose of nitazoxanide (NTZ) within seven days prior to screening.
* Known sensitivity to nitazoxanide (NTZ) or any of the excipients comprising the study medication.
* Subjects unable to swallow oral tablets or capsules.
* Subjects with known severe heart, lung, neurological or other systemic disease that the Investigator believes could preclude safe participation.
* Subjects likely or expected to require hospitalization unrelated to cold during the study period.
* Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol including completion of the subject diary.
* Subjects taking medications considered to be major CYP2C8 substrates.
* Persons with any clinical sign or symptoms suggestive of severe systemic illness with COVID-19, including the following:

  1. shortness of breath at rest,
  2. resting pulse ≥125 beats per minute,
  3. resting respiratory rate ≥ breaths per minute, or
  4. SpO2 ≤ 93% on room air at sea level.
* Subjects known to have a diagnostic test positive for SARS-CoV-2 or influenza infection within the preceding three weeks.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - HealthStar Research LLC, Hot Springs, Arkansas
  - Invesclinic US LLC, Fort Lauderdale, Florida
  - RH Medical Urgent Care, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nitazoxanide | Placebo
Started | 104 | 110
Completed | 101 | 107
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitazoxanide | Placebo | Total
Number analyzed (Participants) | 104 | 110 | 214
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (14.7) | 35 (13.9) | 36 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 74 | 143
  Male | 35 | 36 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 19 | 33
  Not Hispanic or Latino | 90 | 90 | 180
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 13 | 18
  White | 97 | 92 | 189
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 4 | 5
Baseline Illness Severity [Count of Participants; unit: Participants] — Mild illness is defined as baseline assessments of (1) resting pulse <90 beats per minute and (2) resting respiratory rate <20 breaths per minute.
  Moderate illness is defined as baseline assessments of (1) resting pulse ≥90 beats per minute or (2) resting respiratory rate ≥20 breaths per minute.
  Participants
    Mild Illness | 73 | 68 | 141
    Moderate Illness | 31 | 42 | 73
Subject Risk Status [Count of Participants; unit: Participants] — Risk factors for severe illness or complications of EV/RV infection include: Subjects with COPD, Type 2 diabetes mellitus, BMI ≥30, chronic kidney disease, sickle cell disease, serious heart conditions, asthma (moderate or severe), cerebrovascular disease, cystic fibrosis, hypertension or high blood pressure, immunocompromised state, neurologic conditions , liver disease, pulmonary fibrosis, past or present history of smoking, thalassemia, or type 1 diabetes mellitus. Subjects who are ≥65 years of age.
  Participants
    At Increased Risk of Complications | 62 | 67 | 129
    Not At Increased Risk of Complications | 42 | 43 | 85
Time from Symptom Onset to Randomization [Mean (Standard Deviation); unit: hours] | 39 (15.0) | 40 (15.6) | 39 (15.3)

OUTCOME MEASURES:

1. Primary Outcome: Time From First Dose to Sustained Response
Description: Time to Sustained Response is the time in days from the first dose of study medication to the first time at which the subject reports a decrease in total FLU-PRO score from the previous diary with assessment that symptoms are at least "somewhat better than yesterday", no oral temperature ≥100.4 F in the prior 24 hours, and no future increase in any of the FLU-PRO domains except within validated background levels.
  NOTE: Data collection ended at study day 21 and >25% of subjects in each treatment group had not yet achieved Sustained Response (32% in the Nitazoxanide group and 35% in the Placebo group). Therefore, it was impossible to calculate a third quartile for either group. Data presented here imputes "21" as the third quartile. No statistical analyses were performed as enrollment was terminated early. See caveats and limitations.
Time Frame: 21 days
Population: All randomized subjects who received at least one dose of study medication and were positive at Baseline for enterovirus/rhinovirus (EV/RV) infection.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 79 | 92
days | 13.5 [6.22 to 21] | 16.3 [7.32 to 21]

2. Secondary Outcome: Proportion of Subjects Requiring Systemic Antibiotics
Description: Proportion of subjects requiring systemic antibiotics for an infection secondary to Enterovirus/Rhinovirus. NOTE: No statistical analyses were performed as enrollment was terminated early. See caveats and limitations.
Time Frame: 21 days
Population: All randomized subjects who received at least one dose of study medication and were positive at Baseline for enterovirus/rhinovirus (EV/RV) infection. Proportions rounded to the nearest hundredth.
Measure: Number; unit: proportion of participants
Arm/Group | Nitazoxanide | Placebo
Number analyzed (Participants) | 79 | 92
proportion of participants | 0.03 | 0.07

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Nitazoxanide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/110
Other Adverse Events (participants affected / at risk) | 3/104 | 6/110
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitazoxanide (N=104) | Placebo (N=110)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Enrollment was paused due to the COVID-19 pandemic in early 2021 with intention of resuming enrollment at a later date. Ultimately, the study was terminated prior to reaching the enrollment goal. Fewer than half of the planned number of patients were enrolled. Study results are summarized descriptively, but no statistical analyses were performed due to sample size insufficient for statistical comparison.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/81/NCT04489381/Prot_SAP_000.pdf